CLINICAL TRIAL: NCT04391517
Title: Non-invasive Measurement of Serum Haemoglobin in a Perioperative Setting
Brief Title: SpHb Perioperatively
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SpHbv1.2
Record Dates: First submitted 2020-05-02; First posted 2020-05-18 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Anemia; Anemia, Iron Deficiency
Keywords: Patient Blood Management; Perioperative; Anemia
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Population (Experimental): Included patients will be evaluated by an anaesthesiologist according to national and international guidelines as it is routine at the pre-operative clinic. In addition, all included patients will have their Hb measured non-invasively by a trained health care provider. SpHb values will be recorded in the documentation software already in use at the clinic.
  Interventions: Diagnostic Test: SpHb measurement

INTERVENTIONS:
Diagnostic Test: SpHb measurement — All included patients will have their Hb measured non-invasively by a trained health care provider. SpHb values will be recorded in the documentation software already in use at the clinic.

SUMMARY:
This study's goal is to establish SpHb threshold values that can help health care provider sort out which patients would potentially benefit from central laboratory Hb testing pre-operatively and who would likely not. It also aims to compare the mean difference between these two methods in a pre-operative setting.

SpHb values will be observed and recorded from patients meeting the inclusion criteria undergoing pre-operative evaluation for plastic, trauma, orthopaedic, urological, general and gynaecological surgery over one year by the Department of Anaesthesiology and Intensive Care Medicine at the University Medical Centre Graz.

All patients will be evaluated pre-operatively by an anaesthesiologist, utilizing both central laboratory measurements as clinical routine and non-invasive Hb measurements. Both measurements (SpHb and central laboratory Hb) will be documented, along with the normally collected patient data, using the electronic system currently in use. Median values from the two methods will be compared, and possible cut-off values calculated.

DETAILED DESCRIPTION:
Knowledge of patients' serum haemoglobin (Hb) levels is of great importance in many areas of medical practice. Standard methods of measurement require direct blood sampling; they are therefore relatively invasive, costly, and time-consuming.

Non-invasive Hb measurement techniques utilizing a finger probe (SpHb) have attracted a lot of attention over the last five years. Numerous studies have compared the accuracy of these devices with central laboratory Hb data in a wide range of clinical settings: operating rooms, critical care units, emergency departments, and blood donor clinics.

A meta-analysis of previous studies regarding SpHb measurements in perioperative and intensive care settings has revealed a mean difference between non-invasive and central laboratory Hb results of 0.10±1.37 g/dl (n=4425) (2) . To date, however, few studies have assessed the use of these devices in a pre-operative setting.

Such a study could be of great value, as Hb measurement plays an important role in the implementation of PBM programmes (Patient Blood Management), which in turn are associated with improved patient outcomes, fewer transfusions and lower costs.

Various guidelines with the aim of reducing unnecessary testing have been proposed. Such guidelines prioritize the tests to be applied during preparation for minor, intermediate and major surgery, considering specific comorbidities.

This study's goal is to establish SpHb threshold values that can help health care provider sort out which patients would potentially benefit from central laboratory Hb testing pre-operatively and who would likely not. It also aims to compare the mean difference between these two methods in a pre-operative setting.

With reliable cut-off values, SpHb levels could serve as a pre-test for patients with a low ASA (American Society of Anesthesiologists) score undergoing minor to intermediate surgery-i.e., those who would normally not receive a complete lab-test before an operation. This adaptation of clinical routine could help to detect anemia where it might otherwise be missed.

To achieve this goal, SpHb values will be observed and recorded from patients meeting the inclusion criteria undergoing pre-operative evaluation for plastic, trauma, orthopaedic, urological, general and gynaecological surgery over one year by the Department of Anaesthesiology and Intensive Care Medicine at the University Medical Centre Graz.

All patients will be evaluated pre-operatively by an anaesthesiologist, utilizing both central laboratory measurements as clinical routine and non-invasive Hb measurements. Both measurements (SpHb and central laboratory Hb) will be documented, along with the normally collected patient data, using the electronic system currently in use. Median values from the two methods will be compared, and possible cut-off values calculated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient planned for elective surgery
* Patient undergoing pre-operative evaluation by an anaesthesiologist
* Informed consent

Exclusion Criteria:

* Age < 18 years
* Patient refusal
* Emergency surgery
* No central laboratory Hb test available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1284 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
SpHb Accuracy | before surgery
  Accuracy (trueness and precision) of non-invasive Hb measurement
SpHb Cut-off | before surgery
  Potential SpHb cut-offs to reliably non-invasively detect anaemia as defined by the gold-standard

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Honnef, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Landeskrankenhaus Universitätsklinikum Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/17/NCT04391517/Prot_SAP_000.pdf